CLINICAL TRIAL: NCT01352624
Title: Improving Money Management Skills for Veterans With Psychiatric Disabilities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Duke University (Other); Durham VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: H133G100145
Record Dates: First submitted 2011-05-10; First posted 2011-05-12 (Estimated); Last update posted 2018-06-15 (Actual); Status verified 2014-09

CONDITIONS: Psychiatric Problem

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental (Experimental): $teps for Achieving Financial Empowerment ($AFE)
  Interventions: Behavioral: $AFE
- Usual Care (No Intervention): Veterans in control arm will receive usual care at VA

INTERVENTIONS:
Behavioral: $AFE — $teps for Achieving Financial Empowerment ($AFE) is an individualized, psycho-educational intervention that aims to teach veterans with psychiatric disabilities how to save money, create a viable budget, avoid money scams and financial exploitation, and access vocational and mental health resources.
  Arms: Experimental

SUMMARY:
Veterans with psychiatric disabilities face unique challenges concerning money management. Financial strain, money mismanagement, and homelessness have been well documented among veterans with psychiatric disabilities and linked to poor outcomes. The investigators' long-term goal is to promote recovery among veterans with psychiatric disabilities by addressing an 'unmet need' of developing basic money skills necessary for independent functioning in living, working, and social environments. The investigators' objective in the current application is to rigorously evaluate a pilot-tested, stakeholder-informed intervention grounded in principles of psychiatric rehabilitation designed to help develop money management skills and informed financial judgment among veterans with psychiatric disabilities. $teps for Achieving Financial Empowerment ($AFE) is an individualized, psycho-educational intervention that aims to teach veterans with psychiatric disabilities how to save money, create a viable budget, avoid money scams and financial exploitation, and access vocational and mental health resources. To evaluate the $AFE, the investigators will randomly assign N=200 veterans with psychiatric disabilities to either (a) the $AFE intervention (n=100); or (b) a "usual care" control (n=100). The investigators will interview veterans with psychiatric disabilities at baseline and six months. The investigators' central hypothesis, based on strong preliminary data, is that by fostering financial skills and judgment, the $AFE will concurrently increase employment, boost work motivation, and reduce disablement. If these outcomes are met, the investigators hypothesize the intervention will also lead to reduced psychiatric symptoms and homelessness among veterans with psychiatric disabilities.

DETAILED DESCRIPTION:
Veterans with psychiatric disabilities face unique challenges concerning money management. Not only do they encounter problems as do non-veterans with psychiatric disabilities; for example, they may possess limited financial experience due to longstanding dependence on family or have limited money skills related to cognitive deficits. But since veterans can receive disability benefits from both the Veteran's Administration (VA) and the Social Security Administration (SSA), the added income paradoxically exposes veterans to greater risk of severe debt and financial exploitation. To compound this problem, VA and SSA policies for working while disabled differ, often change, and thus can be misunderstood in ways that potentially reduce incentives to seek employment.

Financial strain, money mismanagement, and homelessness have been well documented among veterans with psychiatric disabilities and linked to poor outcomes. Hundreds of thousands of veterans have psychiatric disabilities - a number likely to grow as a substantial proportion of troops return from Iraq and Afghanistan. Yet little systematic research has examined how to help veterans with psychiatric disabilities learn tangible skills needed to maintain financial stability in the community. Our long-term goal is to promote recovery among veterans with psychiatric disabilities by addressing an 'unmet need' of developing basic money skills necessary for independent functioning in living, working, and social environments.

Our objective in the current application is to rigorously evaluate a pilot-tested, stakeholder-informed intervention grounded in principles of psychiatric rehabilitation designed to help develop money management skills and informed financial judgment among veterans with psychiatric disabilities. $teps for Achieving Financial Empowerment ($AFE) is an individualized, psycho-educational intervention that aims to teach veterans with psychiatric disabilities how to save money, create a viable budget, avoid money scams and financial exploitation, and access vocational and mental health resources.

To evaluate the $AFE, the investigators will randomly assign N=200 veterans with psychiatric disabilities to either (a) the $AFE intervention (n=100); or (b) a "usual care" control (n=100). The investigators will interview veterans with psychiatric disabilities at baseline and six months. Our central hypothesis, based on strong preliminary data, is that by fostering financial skills and judgment, the $AFE will concurrently increase employment, boost work motivation, and reduce disablement. If these outcomes are met, the investigators hypothesize the intervention will also lead to reduced psychiatric symptoms and homelessness among veterans with psychiatric disabilities.

The investigators are well prepared to pursue this study because of our peer-reviewed research in this area and success in completing large-scale empirical studies of veterans and non-veterans with psychiatric disabilities. The current research is innovative because it will lead to a brief, targeted, cost-effective, feasible procedure for helping veterans potentially become less reliant on disability funds and more likely to work, gaining independence in the community.

At the end of this project, the investigators expect to show that a systematic, evidence-based approach can greatly bolster self-determination and empowerment for veterans with psychiatric disabilities. The investigators plan to construct a user-friendly, transportable manual so clinicians can readily implement the $AFE intervention. The investigators anticipate the primary impact of this study will be evaluation of a novel and effective method to promote independent living and employment and maximize full society integration among veterans with psychiatric disabilities.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* Veteran
* Receives disability for psychiatric or cognitive condition from either the VA or SSA

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2011-04; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Employment | Past six months
  Any part time or full time employment between baseline interview and follow-up interview

SECONDARY OUTCOMES:
Financial savings | Past Six months
  Amount of money saved between baseline and follow-up interview
Financial Debt | Past six months
  Amount of unsecured debt incurred between baseline and follow-up interviews
Homelessness | Past Six Months
  Homeless and/or living in a homeless shelter for at least one day between baseline and follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Eric Elbogen, Ph.D., Principal Investigator — UNC-Chapel Hill; Eric Elbogen, Ph.D., Principal Investigator — UNC Chapel Hill
Locations (1):
- Duke University, Durham, North Carolina, United States

REFERENCES:
- [Derived] Elbogen EB, Hamer RM, Swanson JW, Swartz MS. A Randomized Clinical Trial of a Money Management Intervention for Veterans With Psychiatric Disabilities. Psychiatr Serv. 2016 Oct 1;67(10):1142-1145. doi: 10.1176/appi.ps.201500203. Epub 2016 May 16. PMID 27181733